CLINICAL TRIAL: NCT01114789
Title: Impact on the Proteolysis of Obesity in Dialysis
Acronym: IPOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Centre Hospitalier de Vichy (Other); AURA Auvergne Dialyse (Association pour l'Utilisation du Rein Artificiel Auvergne) (Unknown)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-0071; 2008-A00729-46 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Hemodialysis Patients
Keywords: chronic renal failure; hemodialysis; obesity; proteolysis
MeSH Terms: conditions — Kidney Failure, Chronic; Obesity | interventions — Proteolysis

INTERVENTIONS:
Other: Proteolysis — protocol designed to examine the effect of obesity on muscle proteolysis in hemodialysis and control

SUMMARY:
The objective of this study is to determine whether obesity has a protective effect on muscle proteolysis in hemodialysis patients submitted to a short starvation. This effect will be tested by comparing measuring muscle proteolysis, using regional infusion of a tracer amino acid (D5 phenylalanine) in two groups of obese and non-obese patients compared to obese and non-obese control subjects.

DETAILED DESCRIPTION:
In hemodialysis patients, the risk of death decreases almost linearly as BMI increases, including in obese patients. Experimental data suggest that obesity may be associated with a reduction of muscle proteolysis during fasting.

In the hemodialysis patients, after an overnight fast an increased use of endogenous energy stores has been reported. The objective of the study is to evaluate the potentially "protective" effect of obesity on protein catabolism during short fasting periods.

Twenty non diabetic patients (men and women) on maintenance hemodialysis for more than six months, aged of 30 to 70 years, will be included: 10 obese (BMI ≥ 30) and 10 non obese patients (18.5 <BMI <25) will be compared with 20 healthy volunteers (men and women) aged 30 to 70 years, obese and non obese, according to the same criteria.

On the investigation day, tracer kinetic studies will be associated with resting energy expenditure measurements and body composition analysis (using dual energy x-ray absorptiometry (DXA).

ELIGIBILITY:
Inclusion Criteria:

* Common Criteria for patients and healthy volunteers:
* Males and females.
* Age between 30 to 70 years.
* Body Mass Index:

Selection criteria for the obese: BMI> 30 kg/m2, Selection criteria for non-obese subjects: 18.5 <BMI <25 kg/m2.

* Biological Review considered satisfactory by the investigator based on the topics covered: chronic renal (obese or not) or healthy volunteers.
* Serology HIV and HCV negative.
* Subject giving his written informed consent
* Affiliated to National Health Insurance

Specific criteria for kidney chronic patients in hemodialysis:

* Patients on hemodialysis since more than 6 months.
* Patients with a clinical stable condition defined by the absence of progressive disease.

Specific criteria for healthy volunteers:

* Subject considered as healthy after clinical examination and medical questionnaire
* Topic willing to be included in the national register of healthy volunteers.

Exclusion Criteria:

* Common Criteria for patients and healthy volunteers:
* Subject under 30 or over 70 years.
* Pregnant or lactating.
* For women of childbearing age: β-hCG assay positive and not have to contraceptives reliable (oral contraceptive, IUD, implant or hormone patch).
* Medical or surgical history (judged by the investigator to be incompatible with the study).
* Diabetics (type 1 or 2).
* Blood donation in the two months preceding the study.
* Special dietary needs (vegetarian, vegan, ...).
* Heavy alcohol consumption (> 2 to 3 glasses per day depending on sex) or presence of an addiction.
* Tobacco significant (> 5 cigarettes / day or equivalent in cigars or pipe tobacco).
* Intense sporting activity (> 5 hours / week).
* Being in exclusion on the National Volunteers Data file
* Subjects deprived of their liberty by judicial or administrative.

Specific criteria for kidney chronic patients in hemodialysis:

* Patients treated with peritoneal dialysis.
* Patients treated with daily hemodialysis.
* Albuminemia <35 g / l and transthyrétinémie <300 mg / l

Specific criteria for healthy volunteers:

* Refusal to be registered on the National Volunteers Data file
* Currently participating or who having got 4500€ in this year before to have participed in another clinical trial

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Fasting muscle protein kinetics will be assessed by the isotope dilution technique using D5 phenylalanine. The isotopic plasma enrichment in phenylalanine will be measured after collection of arterialized and venous blood of the forearm. | 9h to 13h the day of the investigation

SECONDARY OUTCOMES:
Whole-body protein metabolism will be assessed after 13C-leucine infusion in order to determine proteolysis, protein synthesis and protein balance, | 9h to 13h the day of the investigation
Resting energy metabolism will be measured by indirect calorimetry. | 10h to 11h and 12h to 12h40 the day of the investigation
Lipid metabolism will be investigated by measuring the participation of energy substrates to the energy expenditure, determination of plasma free fatty acids and calculation of VLDL synthesis rates (measuring the isotopic enrichment of apo B100). | the day of the investigation

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, PUPH, Principal Investigator — CHU Clermont-Ferrand (CRNH)
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France